CLINICAL TRIAL: NCT01339039
Title: Phase I Study of Plerixafor (AMD3100) and Bevacizumab for Recurrent High-Grade Glioma
Brief Title: Plerixafor (AMD3100) and Bevacizumab for Recurrent High-Grade Glioma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: Patrick Y. Wen, MD (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor-Investigator, Patrick Y. Wen, MD, Disease Center Leader, Center For Neuro-Oncology, Dana-Farber/Brigham and Women's Cancer Center
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10-329; MAMO0909-6 (Other Grant/Funding Number: Genzyme)
Record Dates: First submitted 2011-04-06; First posted 2011-04-20 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: High Grade Glioma: Glioblastoma (GBM); High Grade Glioma: Gliosarcoma; Anaplastic Astrocytoma (AA); Anaplastic Oligodendroglioma (AO); Mixed Anaplastic Oligoastrocytoma (AOA)
Keywords: AMD3100; plerixafor; Mozobil; bevacizumab
MeSH Terms: conditions — Astrocytoma; Oligodendroglioma | interventions — plerixafor; Bevacizumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Part 1 (Experimental): Maximum Tolerated Dose Determination of Plerixafor (3 weeks on, 1 week off) and Bevacizumab (every 2 weeks)
  Interventions: Drug: Plerixafor; Drug: Bevacizumab
- Part 2 (Experimental): Surgical Arm: Safety evaluation of Plerixafor (3 weeks on, 1 week off) and Bevacizumab (every 2 weeks)
  Interventions: Drug: Plerixafor; Drug: Bevacizumab; Procedure: Surgery
- Part 3 (Experimental): Safety and tolerability of Plerixafor (daily) at MTD dose from Part 1 and Bevacizumab (every 2 weeks)
  Interventions: Drug: Plerixafor; Drug: Bevacizumab

INTERVENTIONS:
Drug: Plerixafor — Given subcutaneously once a day for 3 weeks followed by 1 week off (standard 3x3 design); MTD determined in Part 1 will be used as dose in Part 2.
  Other Names: AMD3100; Mozobil
  Arms: Part 1; Part 2
Drug: Plerixafor — Given subcutaneously once daily; MTD determined in Part 1 will be used as dose in Part 3.
  Other Names: AMD3100; Mozobil
  Arms: Part 3
Drug: Bevacizumab — Given intravenously on days 1 and 15 (10 mg/kg) of each 28-day cycle
  Other Names: Avastin
Drug: Plerixafor — Daily administration for 5-9 days prior to surgery
  Other Names: AMD3100; Mozobil
  Arms: Part 2
Procedure: Surgery — After receiving 5-9 days of Plerixafor (AMD3100) monotherapy, patients proceed to surgery. After recovering from surgery, patients will proceed to 28-day post-surgical cycles of therapy (Plerixafor at the MTD established in Part 1, 21 days on / 7 days off; bevacizumab 10 mg/kg on days 1 & 15).
  Arms: Part 2

SUMMARY:
Plerixafor in combination with bevacizumab is a drug combination that may stop cancer cells from growing abnormally. Bevacizumab, also known as Avastin, is FDA approved for use in patients with recurrent glioblastoma and has been studied extensively in other types of solid tumors. Plerixafor, also known as Mozobil, is FDA approved for use in patients with non-Hodgkin's lymphoma and multiple myeloma and has been used in treatment for other cancers. Information from experiments in laboratories suggests that the combination of plerixafor and bevacizumab may help prevent the growth of gliomas.

Part 1: The investigators are looking for the highest dose of plerixafor that can be given safely with bevacizumab (with a 21 days on/7 days off regimen of plerixafor). The investigators will also do blood tests to find out how the body uses and breaks down the drug combination.

Part 2: The investigators are looking to see if plerixafor can get past the blood-brain barrier and into brain tumors. The investigators will also do blood tests to find out how the body uses and breaks down the drug combination.

Part 3: The investigators are looking for for more information re: safety and tolerability of plerixafor in combination with bevacizumab (with a 28 days on/0 days off regimen of plerixafor). The investigators will also do blood tests to find out how the body uses and breaks down the drug combination.

DETAILED DESCRIPTION:
* This study is organized into cycles. Each cycle lasts four weeks (28 days). Cycles occur back to back without a break in between.
* Plerixafor is given as subcutaneous injection (under the skin). The injection should be given at approximately the same time each day (If participants would like the option to administer their Plerixfor in the evening rather than in the morning on non-clinic days, this is a possibility, provided certain conditions are met). The research doctor will specify which days participants should take plerixafor. In general, plerixafor will be given once daily during the first three weeks of every cycle (during part 3, patients will receive plerixafor the last week of each cycle, as well). For the first week (5-7 days) of Cycle 1, the injections will be given in the clinic and the nurses will teach the participant and their spouse/friend/family member how to administer the injections.
* Bevacizumab (10 mg/kg) will be given as an infusion on Days 1 and 15 of each cycle.
* During Part 1 the investigators are looking for the highest dose of the study drug that can be administered safely in combination with bevacizumab so not everyone who participates will receive the same dose of the study drug. The dose given will depend upon on the number of participants who have been enrolled and how well they have tolerated their doses.
* During Part 2, before patient begins their post-surgical cycles of treatment, plerixafor will be administered daily for 5-9 days at the MTD established in Part 1 of the study; patient will continue to surgery; and once recovered from surgery, patient will begin post-surgical cycles of treatment (plerixafor and bevacizumab) at the MTD/regimen established in Part 1 of the study.
* In addition to taking the study medication, participants will have the following tests and procedures done: physical and neurological exam, assessments of the tumor by MRI or CT scan, routine and research blood tests, routine urine tests, pregnancy test (if applicable), ECG, collection of cerebrospinal fluid (CSF) via spinal tap.
* Participants may remain in this research study as long as their tumor is responding or it is determined that receiving further study drugs will not be safe.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of glioblastoma (GBM), gliosarcoma, anaplastic astrocytoma (AA), anaplastic oligodendroglioma (AO), or anaplastic mixed oligoastrocytoma (AOA). Patients are eligible if the original histology was lower-grade glioma.
* Unequivocal progression by MRI or CT
* Patients with recurrence who undergo resection and are left without measurable or evaluable disease are eligible.
* Patients must have recurrent disease and may have had any number of prior relapses (including no prior relapses) on NON-anti-VEGF(R) containing regimens. Relapse is defined as progression following initial therapy. For patients who progressed on a prior anti-VEGF(R) containing regimen including bevacizumab, only one prior relapse on an anti-VEGF(R) containing regimen is allowed.
* 18 years of age or older
* Karnofsky performance status of 60 or greater
* Normal organ and marrow function as outlined in the protocol
* Ability to understand and willingness to sign a written informed consent document.
* Protocol treatment must begin within 5 consecutive days after registration
* Patients enrolled in Part 2 must be willing to undergo surgical resection and have sufficient pre-treatment archival tumor tissue available for molecular analysis
* Women of child-bearing potential must have a negative serum or urine pregnancy test within 72 hours before the start of the investigational product. In addition, female subjects of child-bearing potential and male subjects with partners of child-bearing potential must agree to use an effective means of birth control while on study therapy and for a minimum of 4 months following last plerixafor dose and 6 months following last bevacizumab dose.

Effective birth control includes:

* birth control pills, depot progesterone, or an intrauterine device plus one barrier method;
* or 2 barrier methods. Effective barrier methods are male and female condoms, diaphragms, and spermicides (creams or gels that contain a chemical to kill sperm). Hormonal contraceptive methods are not sufficient, as information about any interaction of plerixafor with hormonal contraceptives is not known.

Exclusion Criteria:

* Patients who have had prior chemotherapy within the past 4 weeks (6 weeks for nitrosoureas or mitomycin C). Patients must be off treatment with Temozolomide for at least 23 days. Patients who received non-cytotoxic drug therapy must be off treatment for at least 2 weeks. For patients enrolling in Part 1 or Part 3 AND who have progressed on a prior bevacizumab-containing regimen, patients may continue treatment with bevacizumab 10 mg/kg monotherapy, with last dose of bevacizumab administered no fewer than 14 days from start of Plerixafor and bevacizumab. For participants enrolling in Part 1 or Part 3 AND who have progressed on a prior anti-VEGF(R) (other than bevacizumab) containing regimen, patients must be off anti-VEGF(R) treatment for at least 28 days before receiving Plerixafor and bevacizumab. For patients enrolled in Part 2 (surgical substudy) AND who have progressed on a prior bevacizumab or other anti-VEGF(R) containing regimen, patients must be off anti-VEGF(R) treatment for at least 28 days prior to surgery.

NOTE: Participants must have recovered to a grade 0 or 1 from any clinically significant toxicity related to prior therapy (with the exception of lymphopenia, which is common after therapy with temozolomide). For any patient who received prior bevacizumab or an anti-VEGF(R) therapy, patient must NOT have discontinued that treatment regimen due to a treatment-related toxicity.

* In order to prevent registering patients with pseudoprogression rather than true disease progression, patients must not have received any form of cranial radiation within 12 weeks of study entry.

NOTE: Patients who have received cranial radiation within 12 weeks of study entry will be allowed to register to trial only if progressive disease is confirmed via biopsy.

* Major surgical procedure (including craniotomy) or significant traumatic injury less than 28 days or those who receive minor surgical procedures (e.g. core biopsy or fine needle aspiration) within 7 days.
* Patients may not be receiving any other investigational agents within the past 28 days.

NOTE: If agent's half-life x 5 is < 28 days, patient may have taken it within the last 28 days, provided at least 5 half-lives have passed since having last taken it.

* Patients who have had prior therapy with CXCR4 inhibitors.
* Patients with one prior relapse on a bevacizumab or an anti-VEGF(R) (i.e. VEGF-trap, vandetanib, cediranib, sunitinib, sorafenib, XL184, etc.) containing regimen are allowed to participate.
* Prior therapy with thalidomide and lenalidomide is allowed.
* Patients who have received prior treatment with implanted radiotherapy or chemotherapy sources such as wafers of polifeprosan 20 with carmustine (e.g. Gliadel wafers).
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to plerixafor or bevacizumab.
* For the first 20 patients to register, no anti-coagulation is allowed; for all subsequent patients screened, patients requiring therapeutic anticoagulation with warfarin at baseline are excluded (however, therapeutic or prophylactic therapy with a low-molecular weight heparin is acceptable).
* Patients must not have a known coagulopathy that increases risk of bleeding or a history of clinically significant hemorrhages in the past.
* Patients whose MRI scan demonstrates intratumoral hemorrhage or peritumoral hemorrhage are not eligible for treatment if deemed significant by the treating physician.
* Patients with gastrointestinal bleeding or any other hemorrhage/bleeding event CTCAE Grade >/= 3 within 30 days prior to study entry.
* Uncontrolled intercurrent illness including but not limited to uncontrolled hypertension, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with greater than 1+ proteinuria on a urine dipstick or equivalent routine laboratory analysis will require further testing with a urine protein to creatinine ratio.
* History of myocardial infarction, unstable angina, stroke, or TIA within 6 months prior to planned Day 1 of dosing
* History of non-healing wounds or ulcers, or bone refractures within 3 months of fracture
* History of abdominal fistula, gastrointestinal perforation, or intraabdominal abscess within 6 months prior to planned Day 1 of dosing
* HIV-positive patients on combination antiretroviral therapy
* Participants with a history of a different malignancy are ineligible except for the following circumstances: Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years AND are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 3 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin.
* Pregnant and breastfeeding women
* Men or women of childbearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up a minimum of 4 months following last Plerixafor dose and 6 months following last bevacizumab dose.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2017-04-08 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) | 9 months
  To determine the maximum tolerated dose (the highest dose combination that causes DLT in no more than 1 of 6 patients) of plerixafor 3 weeks on, 1 week off in combination with bevacizumab (every two weeks) in this patient population.

SECONDARY OUTCOMES:
Safety Evaluation (3 weeks on / 1 week off) - Assessment of the proportion of subjects with different grades of toxicities | 2 years
  To evaluate the safety of plerixafor 3 weeks on, 1 week off in combination with bevacizumab (every 2 weeks) in this patient population. Safety variables will be summarized by descriptive statistics for Parts 1 and 2. To assess the probability of toxicity associated with the treatment, the proportion of subjects with different grades of toxicities will be estimated along with 95% confidence intervals. AEs that occur will be reported for each dose level and for each Part of the study.
Safety and Tolerability (daily plerixafor) - Assessment of the proportion of subjects with different grades of toxicities | 3 years
  To evaluate the safety and tolerability of once daily plerixafor in combination with bevacizumab (every 2 weeks) in this patient population. Safety variables will be summarized by descriptive statistics for Part 3. To assess the probability of toxicity associated with the treatment, the proportion of subjects with different grades of toxicities will be estimated along with 95% confidence intervals. AEs that occur will be reported for each dose level and for each Part of the study.
Determination of Plasma PK Parameters | 2 years
  To determine the plasma pharmacokinetics of plerixafor in patients receiving bevacizumab (every other week). PK parameters will be calculated from each subject's plerixafor plasma concentration versus time data, and summarized by cohort. The following PK parameters will be determined by non-compartmental analysis: Cmax, Tmax, Clast, Tlast, kel, half-life, AUC0-last, AUCinf, CL, and Vd. Additional parameters may be reported depending on the characteristics of the observed plasma concentration profiles.
Exploratory Objective #1 - Preliminary data assessment on anti-tumor efficacy | 3 years
  Exploratory Objective #1 - Preliminary data assessment on the anti-tumor efficacy of plerixafor in combination with bevacizumab in this population. Since efficacy is not the primary objective, the efficacy variables will be summarized descriptively by treatment cohort. Efficacy evaluations will occur every 8 weeks and will consist of imaging and clinical assessment. The rates of response (Complete Response and Complete Response + Partial Response) will be estimated for each dose cohort in Part 1, the MTD (expanded) cohort in Part 1, Part 2, and Part 3.
Exploratory Objective #2 - Investigation of cerebrospinal fluid (CSF) penetration of plerixafor | 3 years
  Plerixafor levels in the cerebrospinal fluid (CSF) will be examined, since despite the potential of plerixafor in inhibiting vasculogenesis and tumor invasion, it is unlikely to be effective unless adequate concentrations can be achieved in the brain.
Exploratory Objective #3 - Investigation of tumor tissue penetration of plerixafor | 3 years
  Tumor tissue of 10 patients with recurrent HGG who require a reoperation (Part 2) will be examined for plerixafor levels and for evidence of pathway inhibition in vivo, since despite the potential of plerixafor in inhibiting vasculogenesis and tumor invasion, it is unlikely to be effective unless adequate concentrations can be achieved in the brain.
Exploratory Objective #4 - Investigation of the correlation of treatment response with laboratory correlates including circulating biomarkers | 3 years
  The goal of the analysis of the biological correlate data is providing an increased understanding of the nature of the response to plerixafor (AMD3100) and bevacizumab and whether blood and tissue biomarkers can assist in predicting response and progression. These studies are exploratory. The nature of the analyses and the strength of the conclusions from these laboratory studies depend not only on the amount of data available, but also on the nature of patient response to therapy. The information will be limited by the small number of patients treated at each dose.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Y. Wen, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts